CLINICAL TRIAL: NCT05220033
Title: Journey Ahead: Enhancing Coping and Communication for Women Diagnosed With Gynecological Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Chief, Behavioral Sciences, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2019002089; 131908 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2021-11-22; First posted 2022-02-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; Endometrial Cancer; Fallopian Tube Cancer; Cervical Cancer; Uterine Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Journey Ahead (Experimental): Experimental: Journey Ahead intervention focusing on coping and communication skill development during the course of 8 sessions and 6 phone calls.
  Interventions: Other: Informational intervention; Other: survey administration

INTERVENTIONS:
Other: Informational intervention — Receive information focusing on coping skills for patients diagnosed with gynecologic cancer
Other: survey administration — Ancillary studies

SUMMARY:
This study looks at how well the Journey Ahead intervention works in improving coping and communication skills in participants with gynecologic cancers.

DETAILED DESCRIPTION:
Primary goals of this project are:

Objective 1: Phase 1: To collect feedback from patients on CCI online and to assess patient's evaluation of CCI online.

Objective 2: Phase 1: To examine the feasibility and acceptability of a CCI online.

Objective 3: Phase 1/2: To collect preliminary data on changes in distress and coping associated with participation in CCI online.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any stage of primary ovarian cancer, primary peritoneal cancer, or primary fallopian tube cancer or experienced a recurrence in the past 5 years;
* Diagnosed with High Grade Stage 2, any grade Stage 3 or higher endometrial cancer or experienced a recurrence in the past 5 years;
* Diagnosed with Stage 2 or higher cervical cancer or experienced a recurrence within the past 5 years;
* Diagnosed with any stage Uterine Cancer (both Sarcoma and carcinosarcoma) or experienced a recurrence in the past 5 years;
* At the time of recruitment the patient has received chemotherapy or radiation in the past 5 years, or is less than 5 years post-cancer surgery;
* At the time of recruitment, a Karnofsky Performance Status of 80 or above or an Eastern Cooperative Oncology Group (ECOG) (80) score of 0 or 1;
* 18 years of age or older;
* English speaking;
* Has internet access, able to view the online intervention sessions and attend telephone or video/telehealth chats to discuss the session content and provide feedback;
* Must give informed consent within 5 years of diagnosis.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms "change" is being assessed | Baseline, two and 6 months post-baseline
  Depressive symptoms will be measures with the Beck Depression inventory which is a 21-item scale which has been widely used in studies incorporating cognitive-behavioral interventions. Calculate score bye summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63.
Psychological distress and well being "change" is being assessed | Baseline, two and 6 months post-baseline
  The MHI-18 has subscales for Psychological Distress (anxiety, depression and loss of behavioral and emotional control) and Well-being. can assess 4 subscales of emotional status like Anxiety, Depression, Behavioral control, and Positive affect. MHI generates one total score. The subscale and total scores range from 0 - 100, with higher scores indicate better mental health
Cancer specific distress "change" is being assessed over the time points | Baseline, two and 6 months post-baseline
  The Impact of Events Scale (IES) (108) is a 21-item self-report measure focusing on intrusive and avoidant ideation related to ovarian cancer and its treatment. Using a 4-point Likert scale, participants rate how true each statement has been for them during the past week (scale range = 0-75).
Quality of life using the Fact-G "change" is being assessed | Baseline, two and 6 months post-baseline
  The Functional Assessment of Cancer Therapy - General (FACT-G) (110) is a widely used measure of QOL. The FACT-G is comprised of 27 questions that assess well-being in four domains: physical (PWB), functional (FWB), social/family (SFWB), and emotional (EWB). PWB assesses the physical symptoms; FWB assesses the degree to which the person can participate and enjoy normal daily activities; SFWB assesses social support and communication, and EWB measures mood and emotional response to illness. The domains are summed

SECONDARY OUTCOMES:
Physical impairment | Baseline, two and 6 months post-baseline
  The 26 item Physical function scale of the CARES measure asks patients to rate physical limitations on a 5-point scale. The mean of all items is calculated.
Coping "change" is being assessed | Baseline, two and 6 months post-baseline
  The acceptance, positive reappraisal, and mental disengagement subscales of the COPE (Carver, Scheier, Weintraub 1989). The scale ranges from 1 = I usually don't do this at all 2 = I usually do this a little bit 3 = I usually do this a medium amount 4 = I usually do this a lot. The scale assess a broad range of coping responses
Emotional Acceptance scale Change | Baseline, two and 6 months post-baseline
  The Emotional Acceptance Scale (Stanton et. al., 2000) will be administered. Thirteen items include statements such as, "I naturally and easily attend to my feelings," "I allow myself to be in touch with my feelings because it is very good for me", and "Knowing they are 'not perfect', I am comfortable with my feelings as they are." Participants indicate percentage of time they believe the statement is true for them ranging from 0 for "never" to 100 for "almost always." The total score is the average for the 13 items (range 0 - 100) and higher scores indicate more emotional acceptance.
Positive emotional expression | Baseline, two and 6 months post-baseline
  Positive emotional expression is a 7 item subscale of the Emotional Expressiveness Questionnaire (King & Emmons, 1990). Items are rated on a 5-point Likert scale with 0 = Never; 1 = Rarely; 2 = Sometimes; 3 = Frequently; 4 = Always. High scores ndicate a tendency to express emotion.
Holding back from sharing concerns | Baseline, two and 6 months post-baseline
  The degree to which the participant holds back from talking about cancer-related concerns with others will be measured by asking participants to rate how much each of 11 common cancer concerns is a concern and how much they hold back from talking to others about this concern. The Investigators adapted this scale from Porter and colleagues (Porter, et. al, 2005). A 13-item scale was used that measures the degree to which participants hold back from family and friends. Participants are asked to rate, on a 6-point scale, the degree to which they hold back from discussing issues of concern with friends and family. Scores are averaged to produce a total score, with higher scores indicating greater holding back
Unsupportive responses from friends and family | Baseline, two and 6 months post-baseline
  The family and friend version of the perceived negative behavior scale (Manne, Pape, & Taylor, 1999) contains critical responses as well as more subtle responses of others. .Cronbach's alphas have ranged from .87 to .94 in the investigators' work with this patient population (Manne et al., 2019)
Psychological flexibility | Baseline, two and 6 months post-baseline
  The 10-item Acceptance and Action Questionnaire-II will be used (AAQ-II) (Bond et. al., 2011) to assess avoidance and willingness to accept undesirable thoughts and feelings while acting in congruence with personal values and goals. a 1 = never true up to 7 = always true. Higher total scores mean less flexibility, while lower total scores mean more flexibility
Hope | Baseline, two and 6 months post-baseline
  The 6-item State Hope Scale (SHS; Snyder, Sympson, Ybasco, Borders, Babyak, & Higgins, 1996) measures agency (belief in one's ability to reach goals) and pathways (belief in one's ability to find routes to reach goals). Individuals rate how true or false each statement (e.g., "I can think of many ways to reach my current goals.") is for them right now on a scale of 1 (Definitely false) to 8 (Definitely true). Total scores range from 6-48 and subscale scores range from 3-24.

OTHER OUTCOMES:
Demographic information | Baseline only
  items assessing age, education, ethnicity, occupation, employment status, income, religious affiliation, marital status and length of significant relationship (baseline only).
Medical information- type of cancer | Baseline, two and 6 months post-baseline
  Chart reviews at baseline will capture type of cancer
Working alliance inventory | Baseline, two and 6 months post-baseline
  The WAI Short Form (WAI-S) is a 12 item inventory rated on a 7-point Likert scale (A. O. Horvath, 1981, 2010). The measure has three alliance subscales: Bond, Task, and Goal.
Medical Outcome- time since diagnosis | Baseline, two and 6 months post-baseline
  Chart reviews at baseline will capture time since diagnosis
Medical Outcome- use of medication for pain, depression, anxiety | Baseline, two and 6 months post-baseline
  Chart reviews at baseline will capture use of medication for pain, depression, anxiety
Medical outcome- cancer treatment history | Baseline, two and 6 months post-baseline
  Chart reviews at baseline will capture cancer treatment history
Medical outcome- sleep disturbance | Baseline, two and 6 months post-baseline
  Chart reviews at baseline will capture sleep disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Manne, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT05220033/ICF_000.pdf